CLINICAL TRIAL: NCT06130683
Title: Single-Cell Sequence Technology Used to Reveal Heterogeneity of Secondary Hyperparathyroidism
Status: Active, not recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Meng Yang, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: 2023-NHLHCRF-YYPPLC-ZR-08
Record Dates: First submitted 2023-11-03; First posted 2023-11-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Parathyroid glands
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Secondary Hyperparathyroidism: Patients who were diagnosed as secondary hyperparathyroidism
  Interventions: Other: Single-cell sequencing
- Primary Hyperparathyroidism: Patients who were diagnosed as primary hyperparathyroidism
  Interventions: Other: Single-cell sequencing
- Normal group: Parathyroid tissue obtained incidentally during other neck surgeries, derived from people without parathyroid disease.
  Interventions: Other: Single-cell sequencing

INTERVENTIONS:
Other: Single-cell sequencing — Single-cell sequencing technology can reveal the gene structure and gene expression status of individual cells, reflecting the heterogeneity between cells.

SUMMARY:
This project intends to select cases that meet the research requirements, take secondary hyperparathyroidism, primary hyperparathyroidism and normal human parathyroid tissue, a total of three groups, 4 cases in each group, through the method of single-cell transcription and sequencing, construct a map of human parathyroid function types, reveal the gene structure and gene expression status of cells, and visualize the expression characteristics, intercellular heterogeneity, and heterogeneity of cell subsets of secondary hyperparathyroid cells in a hierarchical manner, draw a single-cell map, and compare the differences between groups. To explore the pathogenesis of secondary hyperparathyroidism.

Secondary hyperparathyroidism, parathyroid tissue of primary hyperparathyroidism and normal parathyroid tissue obtained by accident were collected, frozen and preserved, frozen tissue thawed, single-cell suspension was prepared and each cell was specifically labeled by the Mozhuo Genomics system, after oil breaking, polymerase chain reaction amplification, reverse transcription to obtain complementary DNA, and a library of complementary DNA that passed quality inspection was constructed to obtain high-quality data of parathyroid cells. Cell Ranger, R Seurat package, and t-SNE dimensionality reduction diagram were used to reduce the dimensionality, cluster, and visualize the data.

In order to construct a single-cell atlas of parathyroid glands, investigators performed cluster analysis of similar cells according to the gene expression profile, and then visualized the data by t-SNE. According to the results of cell clustering, the specific and highly expressed genes in each cell cluster were identified. Cell populations were identified according to the expression of landmark genes, and the differences in cell types and proportions between groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Study participants with a diagnosis of secondary hyperparathyroidism who underwent surgical treatment
* Study participants with a diagnosis of primary hyperparathyroidism who underwent surgical treatment
* Study participants who have obtained informed consent

Exclusion Criteria:

* Other non-secondary hyperparathyroidism conditions such as primary hyperparathyroidism were excluded at the time of inclusion of study participants with essential hyperparathyroidism.
* Other non-primary hyperparathyroid conditions such as secondary hyperparathyroidism were excluded at the time of inclusion of study participants with essential hyperparathyroidism.
* Refusal of informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who undertake surgery for secondary hyperparathyroidism or primary hyperparathyroidism and other neck surgeries in our China-Japan Friendship Hospital
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Construct the single-cell atlas | One year
  A single-cell atlas of normal parathyroid, primary hyperparathyroidism, and secondary hyperparathyroidism was constructed.
  Differential analysis is performed to explore differences in gene expression. Next step is to perform kegg and analyze the pathway information. Cell populations are used to explore changes in cell state during population progression. Quasi-temporal analysis is designed to delineate the dynamic trajectory of cell differentiation and the dynamic process of gene expression. SCENIC is a network for inferring gene co-expression.
  Investigators will use software such as CellRanger and the Seurat package in R word to implement this.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Yang, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China and Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No